CLINICAL TRIAL: NCT02986724
Title: CHRONOS - A Multicenter, Non - Interventional Study to Observe the Safety and Efficacy of Vedolizumab (Entyvio) in Patients With Ulcerative Colitis or Crohn´s Disease That Are Biologic naïve, Observed in Daily Practice in Austria
Brief Title: A Study to Observe the Safety and Efficacy of Vedolizumab in Biologically Naive Participants With Ulcerative Colitis (UC) or Crohn´s Disease (CD)
Acronym: CHRONOS
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4017
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases
Keywords: Drug therapy
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vedolizumab: Bio-naïve participants with UC or CD will be treated with vedolizumab as per local prescriptions from physician in routine medical practice for up to 52 Week. Participants who fail on vedolizumab may be switched during the study to another biologic treatment as prescribed by the physician during routine medical practice for up to 52 Weeks.

SUMMARY:
The purpose of this non-interventional study (NIS) study is to assess further knowledge on the routine use of Entyvio in inflammatory bowel disease therapy, particularly the use in participants with CD and UC naive to biologics.

DETAILED DESCRIPTION:
The drug being tested in this prospective, observational study is called vedolizumab. Vedolizumab (Entyvio) is being used to treat people who have CD or UC. This study will look in the routine use of vedolizumab in inflammatory bowel disease therapy in participants with CD or UC who did not receive a biologic treatment before. The study will enroll approximately 150 participants. All participants enrolled in this will belong to one observational group: Vedolizumab.

Participants taking vedolizumab as per physician's prescription in routine clinical practice will be observed.

This multi-centre trial will be conducted in Austria. The overall time to participate in this study is 2 years. Participant taking vedolizumab in routine clinical practice will make multiple visits to the clinic at Baseline, Week 20 and 52. Once a participant is switched to subsequent biologic treatment upon failing treatment with vedolizumab, the switching date will be considered as new baseline followed by visits at Week 20 and 52.

ELIGIBILITY:
Inclusion Criteria

1 Initiating vedolizumab for moderately to severely active UC or CD. Exclusion Criteria

1. Participant is enrolled in a clinical trial in which treatment for UC or CD is managed through a protocol,
2. Prior treatment with a biologic agent,
3. Any other reason that, in the Investigator's opinion, makes the participant unsuitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Biologically naïve participants with UC or CD undergoing treatment with Vedolizumab (Entyvio) will be evaluated for safety and efficacy.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With UC Achieving Clinical Response Based on Partial Mayo Score | Baseline up to 52 Weeks
  Clinical response is defined as a decrease in the partial Mayo Score of at least 2 points and >=25% from baseline, with an accompanying decrease in rectal bleeding subscore of >=1 point from baseline or absolute rectal bleeding subscore of <=1 point. Mayo score is an instrument designed to measure disease activity of UC. It consists of 3 subscores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease. Outcome measure is planned to be assessed in bio-naive participants who receive vedolizumab treatment.
Percentage of Participants With CD Achieving Clinical Response Based on Harvey-Bradshaw Index (HBI) | Baseline up to 52 Weeks
  Clinical response is defined as a decrease in HBI score of >=3 points from baseline. HBI score is used to measure the disease activity of CD. It consists of clinical parameters: general well-being (0-4, where higher score means lower well being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools, where higher scores indicating more severe disease.
Number of Bio-naïve Participants Reporting One or More Treatment-emergent Adverse Events | Baseline up to 52 Weeks

SECONDARY OUTCOMES:
Percentage of Participants With UC Achieving Clinical Remission Based on Partial Mayo Score | up to 52 weeks from start of another biological therapy
  Clinical remission is defined as a partial Mayo score of <=2 with no individual subscore >1. Mayo score is an instrument designed to measure disease activity of UC. It consists of 3 subscores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease. Outcome measure is planned to be assessed in participants who failed on vedolizumab during the first 52 weeks and will switch to another biological therapy up to 52 weeks.
Percentage of Participants With CD Achieving Clinical Remission Based on Harvey-Bradshaw Index (HBI) | up to 52 weeks from start of another biological therapy
  Clinical remission is defined as total HBI score of <=4 points. HBI score is used to measure the disease activity of CD. It consists of clinical parameters: general well-being (0-4, where higher score means lower well being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools, where higher scores indicating more severe disease. Outcome measure is planned to be assessed in participants who failed on vedolizumab during the first 52 weeks and will switch to another biological therapy up to 52 weeks.
Percentage of Participants With UC Achieving Durable Clinical Response Based on Partial Mayo Score | up to 52 weeks from start of another biological therapy
  Durable clinical response is defined as clinical response at Week 104, where clinical response is defined as a decrease in the partial Mayo Score of at least 2 points and >=25% from baseline, with an accompanying decrease in rectal bleeding subscore of >=1 point from baseline or absolute rectal bleeding subscore of <=1 point. Mayo score is an instrument designed to measure disease activity of UC. It consists of 3 subscores: stool frequency, rectal bleeding, and physician rating of disease activity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease. Outcome measure is planned to be assessed in participants who failed on vedolizumab during the first 52 weeks and will switch to another biological therapy up to 52 weeks.
Percentage of Participants With CD Achieving Durable Clinical Response Based on Harvey-Bradshaw Index (HBI) | up to 52 weeks from start of another biological therapy
  Durable clinical response is defined as clinical response at Week 104, where clinical response is defined as a decrease in HBI score of >=3 points from baseline. HBI score is used to measure the disease activity of CD. It consists of clinical parameters: general well-being (0-4, where higher score means lower well being), abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools, where higher scores indicating more severe disease. Outcome measure is planned to be assessed in participants who failed on vedolizumab during the first 52 weeks and will switch to another biological therapy up to 52 weeks.
Number of Participants who Failed Vedolizumab Therapy Reporting One or More Treatment-emergent Adverse Events | up to 52 weeks from start of another biological therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Innsbruck, Austria

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.